CLINICAL TRIAL: NCT03259451
Title: Effectiveness of Repetitive Transcranial Magnetic Stimulation in the Treatment of Chronic Neuropathic Pain: Retrospective Study on a Cohort of 149 Patients at Rennes University Hospital, From January 2014 to December 2015
Brief Title: Effectiveness of Repetitive Transcranial Magnetic Stimulation in the Treatment of Chronic Neuropathic Pain
Acronym: rTMS-CIC
Status: Withdrawn | Type: Observational
Why Stopped: No recruitment
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3045_rTMS-CIC
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Chronic Neuropathic Pain
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
A retrospective, monocentric, observational, descriptive, open study of a cohort of 149 patients from January 2014 to December 2015

DETAILED DESCRIPTION:
Neuropathic pain is a public health problem because of its prevalence reaching nearly 7% of the general population and the effectiveness of current treatments often remains incomplete: only 30-40% of patients are relieved of 50% of their pain by a pharmacological approach.

As early as the 1990s, stimulation of the motor cortex by implanted electrodes made it possible to successfully treat certain chronic refractory neuropathic pain. In 1995 it was reported that the application of repeated shocks by transcranial magnetic stimulation of the motor cortex could induce an analgesic effect in a patient suffering from neuropathic pain.

This technique has proved its analgesic efficacy after an induction treatment over 5 days, in the context of chronic pain (neuropathic or fibromyalgia), but all the patients are not responders and there is currently, Of predictive criteria for response. It seems important to continue studies on this non-medicinal, non-invasive therapy with no significant adverse effects.

ELIGIBILITY:
Inclusion Criteria:

- patient older than 18 years old with chronic neuropathic pain who are resistant to drug therapy for which treatment with rTMS is indicated between January 2014 and December 2015

Exclusion Criteria:

* Patient less than 18 years old
* Pregnant woman
* Non-neuropathic pain
* Pain <6 months
* Unbalanced epilepsy
* Patient with a contraindication for cerebral MRI (cochlear implant, ocular metallic foreign bodies, patient with a pacemaker, mechanical valve)
* Psychiatric pathology
* Person subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic neuropathic pain
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of rTMS in the treatment of chronic neuropathic pain in a short term | Day 7
  Improvement of pain symptoms by at least 30% on the numerical scale
Evaluation of the efficacy of rTMS in the treatment of chronic neuropathic pain in a short term (≤ 1 month) | Month 1
  Improvement of pain symptoms by at least 30% on the numerical scale

SECONDARY OUTCOMES:
Evaluate the effectiveness of rTMS in the treatment of long-term chronic neuropathic pain (> 6 months) | Month 6
  Persistence of at least 30% improvement in pain symptoms on a numerical scale at the end of the sixth month (M6)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No